CLINICAL TRIAL: NCT03576157
Title: Impact Evaluation of Maternal Health Information Messaging in India
Brief Title: Kilkari Impact Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Oxford Policy Management (Unknown); University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 90075552
Record Dates: First submitted 2018-06-22; First posted 2018-07-03 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Breast Feeding; Family Planning; Essential Newborn Care; Training of Frontline Health Workers
Keywords: mobile health, Pregnant and postpartum women, Frontline health workers, India
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kilkari (Experimental): Pregnant and postpartum women randomized to the Kilkari arm will receive health information messages over their mobile phone during pregnancy and up to 1 year postpartum.
  Interventions: Other: Kilkari
- Comparison (No Intervention): Existing standard of care; no new health messages

INTERVENTIONS:
Other: Kilkari — Kilkari is an outbound service that delivers weekly, time-appropriate audio messages about pregnancy, childbirth, and childcare directly to families on their mobile phones, starting from the second trimester of pregnancy until the child is one-year-old.
  Arms: Kilkari

SUMMARY:
British Broadcasting Corporation (BBC) Media Action is presently implementing two large scale mobile health (mHealth) initiatives in India: Kilkari and Mobile Academy. Kilkari is an outbound service that delivers weekly, time-appropriate audio messages about pregnancy, childbirth, and childcare directly to families on their mobile phones, starting from the second trimester of pregnancy until the child is one-year-old. Mobile Academy (MA) is an Interactive Voice Response (IVR) in-service audio training course for Accredited social health activists (ASHAs) in India designed to refresh their knowledge of life-saving preventative health behaviors and improve their interpersonal communications skills. Both programs were initiated in Bihar in 2012, and have been scaled widely in a number of states with support from Ministry of Health and Family Welfare (MOHFW) at the national level, National Health Missions (NHM) at the state level, and an alliance of donors (Gates Foundation, USAID, Barr Foundation, and UK Department for International Development (UKAid)).

The Johns Hopkins School of Public Health, Oxford Policy Management, and University of Cape Town are supporting BBC Media Action and the Ministry of Health and Family Welfare (MOHFW) are conducting an external evaluation of both Kilkari and Mobile Academy (MA). The evaluation spans through April 2020.

DETAILED DESCRIPTION:
The Johns Hopkins Global mHealth Initiative, Oxford Policy Management, and University of Cape Town proposes supporting BBC Media Action and the Ministry of Health and Family Welfare (MOHFW) to conduct an external evaluation of Mobile Academy (MA) and Kilkari. In the below text, we outline 6 proposed activities which comprise the evaluation, which are planned from mid 2018 to April 2020.

These studies will help inform program modification and scale-up plans, and will help better understand the effects of maternal mobile messaging in India and globally.

1. Secondary analysis of cross-site trends in key performance indicators (Duration: throughout study):

   Mobile Academy (MA): We will use system generated data to estimate the proportion of ASHAs who have completed MA training across 12 states. We will additionally aim to understand linkages between ASHA's exposure to the MA training content and performance on MA knowledge assessments.

   Kilkari: We estimate that Kilkari users will have differing levels of exposure to the program. For example, some women may not be present when the Kilkari calls come and thus miss out on key content. Analyses of system generated data will aim to measure exposure to Kilkari messages by content area (e.g. nutrition, family planning, etc) across 12 states where implementation has occurred to date. As part of this analysis we'll seek to understand reasons why calls are not received, including phones being out of network, changes in SIM cards, etc.
2. Summative evaluation of Kilkari (Period: April 2018 to December 2019) Objective: To determine the effectiveness of mobile maternal health information messages on key health outcomes in 4 districts of Madhya Pradesh (MP).

   This objective will be carried out through an individually randomized controlled trial initiated in early 2018. We propose conducting household surveys in all 4 study districts among the cohort of women identified during conception, starting in March 2018. Women identified within the 5-7 month of their pregnancy, who have access to a mobile phone, and consent to participate will be interviewed as part of baseline survey and recruited for participation into Kilkari by 8 months of conception (this is intended to mirror timings observed in Kilkari outreach in other states). Among individuals not randomized to receive messages, we would propose delaying implementation for Kilkari for a 12-month window to allow for evaluation activities to take place and additionally glean information which is anticipated to improve the efficiency of implementation / rollout in other areas.
3. ASHA Survey Objective: Identify factors underpinning differences Reproductive Maternal Newborn and Child Health (RMNCH) knowledge and motivation among frontline health workers, including exposure to the Mobile Academy training program.

   As part of the baseline surveys described under activity 2 in MP, we will conduct face to face interviews with all ASHAs (n=1,200) across the four study districts in MP. A sub-sample will also be contacted for a follow-on phone survey a week later, to pilot modules and validate a phone survey tool on knowledge and motivation, which can then be applied to other ASHAs to measure key outcomes as part of MA deployments in other states, including Rajasthan.
4. Post-natal care phone survey Objective: Measure respectful maternity care (RMC) during childbirth, essential newborn care, and infant feeding practices within 0-3 months postpartum As part of baseline survey activities in MP, we propose additionally identifying women in 1-2 districts who are 0 to 3 months postpartum (n=880). Face to face interviews with postpartum women will provide a forum to measure key infant feeding and essential newborn care outcomes. Phone surveys, a week later, with a subset will help develop a validated phone survey tool for their measurement amongst individuals enrolled into Kilkari.
5. Qualitative interviews of both Kilkari and MA in MP and Rajasthan

   Objectives:

   Mobile Academy

   • Understand stakeholder (ASHA, ASHA supervisor and beneficiary) perceptions of MA, including barriers / facilitators underpinning uptake and completion of MA training and enacting its content, and how it affects interpersonal communication between stakeholders.

   Kilkari
   * Understand stakeholder (ASHA, ASHA supervisor and beneficiary) perceptions of Kilkari, including different message content areas, barriers / facilitators to the adoption of Kilkari's recommended RMNCH practices and careseeking behaviors
   * Identify barriers / facilitators for pregnancy and birth registration

   The qualitative research component will complement the summative evaluation and secondary data analysis components. Qualitative research will include in-depth interviews and focus group discussions in both MP and Rajasthan. Differentials in uptake of MA across these settings provides a unique opportunity to understand the characteristics of ASHAs and the larger health systems environment which contribute to MA completion. Among Kilkari beneficiaries, qualitative research can help better understand user perception of content, the extent and mechanism of impact of the messages on health-related knowledge, behavior and relationships.
6. Economic evaluation of Kilkari Objective: To determine the incremental cost-effectiveness of Kilkari as compared to a null scenario of no messages To estimate the value for money of Kilkari, we will estimate the costs of program to all key stakeholders involved-including BBC Media Action, MOHFW, and end-users. To estimate the effects of the program on health outcomes, we will draw from household survey data at baseline and endline amongst individuals exposed and not exposed to messages. Data on changes in careseeking for antenatal care as well the adoption of practices around breastfeeding and family planning will be inputted into the Lives Saved Tool to generate a measure of lives saved associated with program activities. Lives saved will be used to yield an estimate of the incremental Disability-Adjusted Life Years (DALY) averted and ultimately a cost per DALY averted.

ELIGIBILITY:
Inclusion Criteria:

15-45 years 5-7 months pregnant Resident of study area Consents to participation Access to a mobile phone during morning and afternoon

Exclusion Criteria:

<15 years of age Not female Not a resident of study area <5 months and >8 months pregnant Not a Hindi speaker Access to a mobile phone only during the night

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Women 5-7 months pregnant
Enrollment: 5095 (Actual)
Dates: Start 2018-07-07 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding | 0-6 months following delivery
  The study aims to detect a 5% change in the proportion of women who report practicing exclusive breastfeeding
Immediate breastfeeding | 1 hour following delivery
  The study aims to detect a 5% change in the proportion of women who report practicing immediate breastfeeding

CONTACTS AND LOCATIONS:
Overall Officials: Amnesty E LeFevre, PhD, Principal Investigator — Johns Hopkins School of Public Health, University of Cape Town
Locations (2):
- India (2):
  - N/A-- recruitment occurring at household / community level in 4 districts: Rewa, Rajgarh, Mandsaur, Hoshangabad, Rewa, Madhya Pradesh
  - BBC Media Action, Delhi

IPD SHARING:
Plan to Share IPD: No
De-identified data may be made available upon request to study investigators following the publication of study findings.

REFERENCES:
- [Derived] LeFevre AE, Mendiratta J, Jo Y, Chamberlain S, Ummer O, Miller M, Scott K, Shah N, Chakraborty A, Godfrey A, Dutt P, Mohan D. Cost-effectiveness of a direct to beneficiary mobile communication programme in improving reproductive and child health outcomes in India. BMJ Glob Health. 2023 Mar;6(Suppl 5):e009553. doi: 10.1136/bmjgh-2022-009553. PMID 36958740
- [Derived] Bashingwa JJH, Mohan D, Chamberlain S, Scott K, Ummer O, Godfrey A, Mulder N, Moodley D, LeFevre AE. Can we design the next generation of digital health communication programs by leveraging the power of artificial intelligence to segment target audiences, bolster impact and deliver differentiated services? A machine learning analysis of survey data from rural India. BMJ Open. 2023 Mar 17;13(3):e063354. doi: 10.1136/bmjopen-2022-063354. PMID 36931682
- [Derived] LeFevre AE, Shah N, Scott K, Chamberlain S, Ummer O, Bashingwa JJH, Chakraborty A, Godfrey A, Dutt P, Ved R, Mohan D; Kilkari Impact Evaluation Team. The impact of a direct to beneficiary mobile communication program on reproductive and child health outcomes: a randomised controlled trial in India. BMJ Glob Health. 2022 Jul;6(Suppl 5):e008838. doi: 10.1136/bmjgh-2022-008838. PMID 35835477
- [Derived] Ng A, Mohan D, Shah N, Scott K, Ummer O, Chamberlain S, Bhatnagar A, Dhar D, Agarwal S, Ved R, LeFevre AE; Kilkari Impact Evaluation Team. Assessing the reliability of phone surveys to measure reproductive, maternal and child health knowledge among pregnant women in rural India: a feasibility study. BMJ Open. 2022 Mar 10;12(3):e056076. doi: 10.1136/bmjopen-2021-056076. PMID 35273055
- [Derived] Chakraborty A, Mohan D, Scott K, Sahore A, Shah N, Kumar N, Ummer O, Bashingwa JJH, Chamberlain S, Dutt P, Godfrey A, LeFevre AE; Kilkari Impact Evaluation Team. Does exposure to health information through mobile phones increase immunisation knowledge, completeness and timeliness in rural India? BMJ Glob Health. 2021 Jul;6(Suppl 5):e005489. doi: 10.1136/bmjgh-2021-005489. PMID 34312153
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276
- [Derived] LeFevre A, Agarwal S, Chamberlain S, Scott K, Godfrey A, Chandra R, Singh A, Shah N, Dhar D, Labrique A, Bhatnagar A, Mohan D. Are stage-based health information messages effective and good value for money in improving maternal newborn and child health outcomes in India? Protocol for an individually randomized controlled trial. Trials. 2019 May 15;20(1):272. doi: 10.1186/s13063-019-3369-5. PMID 31092278